CLINICAL TRIAL: NCT00013871
Title: Evaluation of the Immunogenicity of Pneumococcal Conjugate Vaccine and Routine Pediatric Immunizations in HIV-Infected Children Treated With Highly Active Antiretroviral Therapy (HAART)
Brief Title: Pneumococcal Vaccine and Routine Pediatric Immunizations in HIV-Infected Children Receiving Anti-HIV Drugs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Purpose: Prevention
Other Study IDs: P1024; PACTG 1024; 10609 (Registry Identifier: DAIDS ES Registry Number); ACTG P1024
Record Dates: First submitted 2001-03-31; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Hepatitis B; Measles; Pneumococcal Infections; Pertussis
Keywords: Measles-Mumps-Rubella Vaccine; Antibodies, Viral; Hepatitis B Vaccines; Immunization, Secondary; Pneumococcal Vaccines; Antiretroviral Therapy, Highly Active; Diphtheria-Tetanus-acellular Pertussis Vaccines
MeSH Terms: conditions — HIV Infections; Hepatitis B; Measles; Pneumococcal Infections; Whooping Cough; Neoplasm Metastasis | interventions — Tetanus Toxoid; Measles-Mumps-Rubella Vaccine; Pneumococcal Vaccines; Heptavalent Pneumococcal Conjugate Vaccine; Hepatitis B Vaccines

INTERVENTIONS:
Biological: Diphtheria & Tetanus Toxoids & Acellular Pertussis Vaccine Adsorbed
Biological: Measles-Mumps-Rubella Vaccine (Live)
Biological: Pneumococcal Vaccine, Polyvalent (23-valent)
Biological: Pneumococcal Conjugate Vaccine, Heptavalent
Biological: Hepatitis B Vaccine (Recombinant)

SUMMARY:
The purpose of this study is to determine if 2 doses of Pneumococcal Conjugate Vaccine (PCV) followed by 1 dose of Pneumococcal Polysaccharide Vaccine (PPV) in HIV-infected children on anti-HIV therapy is helpful and safe in fighting pneumococcal infections in this group of children. This study will also look at the protection provided by childhood vaccination against measles, pertussis, and hepatitis B virus.

Pneumococcal infections are the most common AIDS-related infection in HIV-infected children. PCV may help reduce the chances of HIV-infected children getting pneumococcal infections. This study will look at whether pneumococcal vaccines are safe and effective in HIV-infected children receiving HAART. It will look at whether HIV-infected children are protected by childhood vaccines received previously and if more doses are safe and improve protection.

DETAILED DESCRIPTION:
Infection by Streptococcus pneumoniae is the most frequent opportunistic infection observed in HIV-infected children. PCVs are immunogenic and efficacious in normal children and offer hope of reducing pneumococcal infections in HIV-infected children. The degree to which children on HAART are protected by prior immunizations and are responsive to new immunizations is still largely undefined. This study is designed to answer whether PCV immunizations are safe and effective. The immune responses to prior immunizations and responsiveness to booster doses of vaccines against measles, pertussis, and hepatitis B virus of children on HAART will also be examined. Answers to these questions will determine whether these children are likely to be protected against these clinically relevant pathogens and whether they should routinely receive booster doses of these vaccines after a period of HAART.

Patients are stratified on the basis of CD4 percentage and age. Patients that previously received a primary hepatitis B vaccine (HBV) series receive an HBV immunization at entry. Other vaccinations may be given (based on age and/or CD4 cell measurement, and immunization status) for PCV at entry and 2 months, and measles-mumps-rubella (MMR) vaccine and PPV at 4 months. Some patients may be administered DTaP at a 6-month visit on the basis of age, previous immunization history, and negative tetanus antibody status. Follow-up visits are done at 8, 12, and 24 months. Blood samples are collected at all clinic visits for assessment of HIV RNA, immune responses against pneumococcus, measles, pertussis, and hepatitis B virus, as well as for laboratory evaluations.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are 2 to 18 years of age.
* Are HIV-infected.
* Have a viral load (amount of HIV in the blood) under 60,000 copies/ml within 30 days of study entry.
* Have been on their current anti-HIV drugs for at least 3 months.
* Have received 4 or more doses of a pertussis vaccine.
* Have received 1 or more doses of measles vaccine unless a CD4 percent or CD4 number ruled out taking the vaccine. (This reflects a change in the CD4 requirement.)
* Expect to be able to complete all study injections and follow-up.
* Have a negative pregnancy test if able to have children and use effective methods of birth control.
* Have parent or guardian's consent if under 18 years of age.
* Have received an approved hepatitis B vaccine series. Not required for study entry, but children who have received this vaccine will be studied.
* (This study was changed to allow patients who became HIV infected after birth, have a viral load between 30,000 and 60,000 copies/ml, and who have been on their current anti-HIV drugs for 3 to 6 months.)

Exclusion Criteria

Patients will not be eligible for this study if they:

* Had a certain CD4 level before beginning anti-HIV drugs and at screening.
* Have received any killed vaccine within 4 weeks, or any live vaccine within 6 weeks, of entering the study.
* Have received pneumococcal vaccines or had a reaction to PPV.
* Have had an allergic reaction to any measles or hepatitis B vaccines, or to other routine childhood immunizations if 13 years of age or less.
* Have any other condition that would make receiving study vaccines inadvisable.
* Are currently on medications that affect the immune system, except for G-CSF and erythropoietin. This includes the equivalent to more than 1 mg/kg/day of prednisone in the 2 weeks preceding study screening. Nonsteroidal anti-inflammatory agents and inhaled corticosteroids are not excluded.
* Have received certain blood products within the previous 6 months.
* Have other diseases of the immune system.
* Have had cancer within 3 months of study screening or are being treated or have been treated for cancer within 3 months of study entry.
* Are pregnant.
* Have any other disease or previous surgery that would interfere with study treatment.
* Are likely to have bleeding disorders.
* Show certain side effects to vaccines at screening.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300
Dates: Study Completion 2004-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Abzug, Study Chair
Locations (40):
- United States (38):
  - UAB, Dept. of Ped., Div. of Infectious Diseases, Birmingham, Alabama
  - Long Beach Memorial Med. Ctr., Miller Children's Hosp., Long Beach, California
  - Usc La Nichd Crs, Los Angeles, California
  - Children's Hosp. & Research Ctr. Oakland, Ped. Clinical Research Ctr. & Research Lab., Oakland, California
  - UCSD Mother-Child-Adolescent Program CRS, San Diego, California
  - UCSF Pediatric AIDS CRS, San Francisco, California
  - Univ. of Colorado Denver NICHD CRS, Aurora, Colorado
  - Connecticut Children's Med. Ctr., Hartford, Connecticut
  - Yale Univ. School of Medicine - Dept. of Peds., Div. of Infectious Disease, New Haven, Connecticut
  - Children's National Med. Ctr. Washington DC NICHD CRS, Washington D.C., District of Columbia
  - South Florida CDTC Ft Lauderdale NICHD CRS, Fort Lauderdale, Florida
  - Univ. of Florida College of Medicine-Dept of Peds, Div. of Immunology, Infectious Diseases & Allergy, Gainesville, Florida
  - Univ. of Florida Jacksonville NICHD CRS, Jacksonville, Florida
  - Univ. of Miami Ped. Perinatal HIV/AIDS CRS, Miami, Florida
  - Columbus Regional HealthCare System, The Med. Ctr., Columbus, Georgia
  - Univ. of Chicago - Dept. of Peds., Div. of Infectious Disease, Chicago, Illinois
  - Chicago Children's CRS, Chicago, Illinois
  - Univ. of Maryland Med. Ctr., Div. of Ped. Immunology & Rheumatology, Baltimore, Maryland
  - Johns Hopkins Hosp. & Health System - Dept. of Peds., Div. of Infectious Diseases, Baltimore, Maryland
  - HMS - Children's Hosp. Boston, Div. of Infectious Diseases, Boston, Massachusetts
  - BMC, Div. of Ped Infectious Diseases, Boston, Massachusetts
  - Baystate Health, Baystate Med. Ctr., Springfield, Massachusetts
  - WNE Maternal Pediatric Adolescent AIDS CRS, Worcester, Massachusetts
  - Rutgers - New Jersey Medical School CRS, Newark, New Jersey
  - SUNY Downstate Med. Ctr., Children's Hosp. at Downstate NICHD CRS, Brooklyn, New York
  - Schneider Children's Hosp., Div. of Infectious Diseases, New Hyde Park, New York
  - Nyu Ny Nichd Crs, New York, New York
  - Columbia IMPAACT CRS, New York, New York
  - Harlem Hosp. Ctr. NY NICHD CRS, New York, New York
  - Cornell Univ., Div. of Ped. Infectious Diseases & Immunology, New York, New York
  - Metropolitan Hosp. Ctr., New York, New York
  - St. Luke's-Roosevelt Hosp. Ctr., New York, New York
  - Strong Memorial Hospital Rochester NY NICHD CRS, Rochester, New York
  - SUNY Stony Brook NICHD CRS, Stony Brook, New York
  - Bronx-Lebanon Hosp. IMPAACT CRS, The Bronx, New York
  - Montefiore Med. Ctr. - AECOM, The Bronx, New York
  - St. Christopher's Hosp. for Children, Philadelphia, Pennsylvania
  - Texas Children's Hosp. CRS, Houston, Texas
- Puerto Rico (2):
  - San Juan City Hosp. PR NICHD CRS, San Juan
  - Univ. of Puerto Rico Ped. HIV/AIDS Research Program CRS, San Juan

REFERENCES:
- [Derived] Abzug MJ, Qin M, Levin MJ, Fenton T, Beeler JA, Bellini WJ, Audet S, Sowers SB, Borkowsky W, Nachman SA, Pelton SI, Rosenblatt HM; International Maternal Pediatric Adolescent AIDS Clinical Trials Group P1024 and P1061s Protocol Teams. Immunogenicity, immunologic memory, and safety following measles revaccination in HIV-infected children receiving highly active antiretroviral therapy. J Infect Dis. 2012 Aug 15;206(4):512-22. doi: 10.1093/infdis/jis386. Epub 2012 Jun 12. PMID 22693229
- [Derived] Abzug MJ, Warshaw M, Rosenblatt HM, Levin MJ, Nachman SA, Pelton SI, Borkowsky W, Fenton T; International Maternal Pediatric Adolescent AIDS Clinical Trials Group P1024 and P1061s Protocol Teams. Immunogenicity and immunologic memory after hepatitis B virus booster vaccination in HIV-infected children receiving highly active antiretroviral therapy. J Infect Dis. 2009 Sep 15;200(6):935-46. doi: 10.1086/605448. PMID 19663708
- [Derived] Abzug MJ, Song LY, Fenton T, Nachman SA, Levin MJ, Rosenblatt HM, Pelton SI, Borkowsky W, Edwards KM, Peters J; International Maternal Pediatric Adolescent AIDS Clinical Trials Group P1024 Protocol Team. Pertussis booster vaccination in HIV-infected children receiving highly active antiretroviral therapy. Pediatrics. 2007 Nov;120(5):e1190-202. doi: 10.1542/peds.2007-0729. Epub 2007 Oct 15. PMID 17938165